CLINICAL TRIAL: NCT00261209
Title: Study of Collagenase Injection Therapy for Treatment of Zone II Flexor Tendon Adhesions in the Hand
Brief Title: Collagenase in the Treatment of Zone II Flexor Tendon Adhesions in the Hand
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Marie A. Badalamente, Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tendon 101
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Adhesion of Flexor Tendon of Hand
Keywords: Flexor Tendon Adhesions; Zone II of the Hand
MeSH Terms: interventions — Collagenases; Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Collagenase Injection (Experimental): Injection of collagenase into adhesion restricting tendon gliding
  Interventions: Drug: Collagenase; Drug: Collagenase injection

INTERVENTIONS:
Drug: Collagenase — Collagenase injection into adhesion restricting tendon gliding
  Other Names: Collagenase Clostridium Histolyticum
Drug: Collagenase injection — injection of collagenase into adhesion restricting tendon gliding
  Other Names: Collagenase Clostridium Histolyticum

SUMMARY:
The purpose of this study is to dissolve flexor tendon adhesions associated with failed tendon repair surgery.

DETAILED DESCRIPTION:
In an open label study, collagenase injection therapy was investigated in 3 subjects for it's ability to lyse flexor tendon adhesions in zone II of the hand.

Results indicate that two of three subjects had improved range of finger motion at the PIP and DIP joints. This may obviate the need for patients to have tenolysis hand surgery to correct the finger flexion contracture of the PIP and DIP joints. Detailed controlled studies remain to be done.

ELIGIBILITY:
Inclusion Criteria:

* zone II flexor tendon adhesion of at least one finger

Exclusion Criteria:

* any chronic, serious or uncontrolled medical condition
* inability to conform to study visits (12-15 per year)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Restoration of PIP and DIP joint motion. | 6 months

SECONDARY OUTCOMES:
Hand Grip strength (kg) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Badalamente, PhD, Principal Investigator — Dept. Orthopaedics, SUNY@Stony Brook, NY 11794; Edward Wang, MD, Principal Investigator — Dept. Orthopaedics, SUNY@Stony Brook, NY 11794
Locations (1):
- Dept. Orthopaedics, SUNY@Stony Brook, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No